CLINICAL TRIAL: NCT00509379
Title: A Phase II Multicenter Non-randomized Study to Assess Safety, Toxicity and Clinical Activity of the Association of Bortezomib(VELCADE)With Rituximab in Relapsed/Refractory Indolent Non Follicular and Mantle-cell Non-Hodgkin Lymphoma
Brief Title: Non-randomized Safety Study With Bortezomib/Rituximab in Relapsed/Refractory Indolent Lymphoma
Acronym: LYM-2023
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano Multiregionale per lo studio dei Linfomi e delle Leucemie (Other)
Collaborators: Centro di Riferimento per l'Epidemiologia e la Prev. Oncologica Piemonte (Other); Fondazione Italiana Linfomi - ETS (Other); University of Turin, Italy (Other)
Responsible Party: Dr. Umberto Vitolo, GIMURELL Onlus
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRIL06; LYM-2023
Record Dates: First submitted 2007-07-30; First posted 2007-07-31 (Estimated); Last update posted 2011-01-28 (Estimated); Status verified 2009-07

CONDITIONS: Lymphoma; Non-Hodgkin Lymphoma
Keywords: Relapsed/refractory indolent lymphoma; Non-follicular Lymphoma; Mantle cell non-Hodgkin Lymphoma; Patients naïve or sensitive to rituximab; Patients not eligible for high dose chemotherapy with ASCT
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin; Recurrence | interventions — Rituximab; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): All patients will be treated with six courses of therapy with a thirteen day rest period between them. Courses will be restarted at day 36.
  Interventions: Drug: Rituximab; Drug: VELCADE

INTERVENTIONS:
Drug: Rituximab — Rituximab 375 mg/m2 as slow iv infusion day 1-8-15-22.Patients will be treated with six courses of therapy with a thirteen day rest period between them. Courses will be restarted at day 36.
Drug: VELCADE — VELCADE 1,6 mg/m2 iv bolus days 1-8-15-22 (Velcade will be administrated prior of Rituximab infusion).Patients will be treated with six courses of therapy with a thirteen day rest period between them. Courses will be restarted at day 36.

SUMMARY:
The promising activity of Bortezomib as single agent in low grade lymphoma patients in small studies has led to a number of larger multicenter trials with Bortezomib in combination with Rituximab in mantle-cell lymphoma, follicular lymphoma and marginal zone lymphoma.

DETAILED DESCRIPTION:
This is a open label, non randomized, phase II , multicenter, prospective trial to evaluate the efficacy and safety of the combination of bortezomib and rituximab in patients with relapsed or refractory rituximab naïve or sensitive indolent non-follicular and mantle cell non-Hodgkin's lymphoma. Despite of the availability of treatment for this disease, this study is justified because no known therapies are really curative and it is necessary to look for new treatment options to improve the clinical outcome and prognosis of relapsed indolent lymphoma. This study is designed for patients not eligible for high-dose chemotherapy and autologous stem cells transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with naïve or sensitive rituximab indolent non-follicular and mantle cell non-Hodgkin's Lymphoma disease that had failed to respond or relapsed after primary therapy. There is a demonstrated progressive disease requiring further treatment. Histological subtype included into the study are are as follows Small lymphocytic/lymphoplasmocytic lymphoma; Nodal marginal zone Lymphoma (MALT lymphoma are excluded) Splenic marginal zone lymphoma Mantle cell lymphoma A lymphnode biopsy is advisable if it is not harmful for the patients, before enrollment of the patient into the study in order to confirm diagnosis and to rule out histologic transformation. Lymphnode biopsy should be performed within 6 months before study entry.
2. Age >18-75
3. Relapse or failure to respond after one or more (maximum three) lines of chemotherapy
4. Any type of prior chemotherapy, rituximab included. Patients who had received high dose chemotherapy and ASCT can be enrolled into the study
5. Naïve or sensitive rituximab disease. If the patient received Rituximab, he/she must have responded and the TTP from the last dose to rituximab must have been 6 months or more.
6. Measurable and/or evaluable disease.
7. Adequate haematological counts: ANC> 1.0 x 109/L and PLT counts> 75 x 109/L unless due to bone marrow involvement by lymphoma.
8. Conjugated bilirubin up to 2 x ULN.
9. Alkaline phosphatase and transaminases up to 2 x ULN.
10. Creatinine clearances> 30 m/min.
11. Non peripheral neuropathy or CNS disease.
12. Life expectancy> 6 months.
13. Performance status< 2 according to ECOG scale.
14. Written informed Consent

Exclusion Criteria:

1. Has known or suspected hypersensitivity or intolerance to rituximab, boron, mannitol, or heparin, if an indwelling catheter is used
2. History of clinically relevant liver or renal insufficiency; significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, rheumatologic, hematologic, psychiatric, or metabolic disturbances
3. Uncontrolled diabetes (if receiving antidiabetic agents, subjects must be on a stable dose for at least 3 months before first dose of study drug
4. Uncontrolled or severe cardiovascular disease including myocardial infarction within 6 months of enrollment, New York Heart Association (NYHA) Class III or IV heart failure (Attachment 5, NYHA Classification of Cardiac Disease), uncontrolled angina, clinically significant pericardial disease, or cardiac amyloidosis
5. History of hypotension or has decreased blood pressure (sitting systolic blood pressure SBP 100 mmHg and/or sitting diastolic blood pressure DBP 60 mmHg)
6. Pregnant or breastfeeding
7. Peripheral Neuropathy or Neuropathic Pain Grade 2
8. HIV positivity
9. HBV positivity with the exception of patients with HBVcAb +, HbsAg -, HBs Ab+/- with HBV-DNA negative
10. HCV positivity with the exception of patients with no signs of active chronic hepatitis histologically confirmed
11. Active opportunistic infection
12. Receipt of extensive radiation therapy, systemic chemotherapy, or other antineoplastic therapy within 4 weeks before enrollment
13. Exposure to Rituximab within 24 weeks before screening
14. Have received an experimental drug or used an experimental medical device within 4 weeks before the planned start of treatment. Concurrent participation in non-treatment studies is allowed, if it will not interfere with participation in this study.
15. Any other co-existing medical or psychological condition that would preclude participation in the study or compromise ability to give informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2006-09; Primary Completion 2007-11 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
To demonstrate a statistical benefit in overall response rate (ORR) of the Bortezomib/Rituximab association in this study 3/13 or fewer responses are observed during the first stage then the trail is stopped early | 1 year

SECONDARY OUTCOMES:
If 12/43 or fewer responses are observed by the end of the trail, then no further investigation of this regimen is warranted | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Umberto Vitolo, MD, Principal Investigator — S.C. Ematologia 2 ASO San Giovanni Battista Torino
Locations (22):
- Italy (22):
  - Ospedale Cardinale Panico, Tricase, Lecce
  - Istituto Clinico Humanitas, Rozzano, Milano
  - Istituto per la ricerca e la cura del cancro, Candiolo, Torino
  - Ospedale Civico, Chivasso, Torino
  - Stabilimento Ospedaliero, Cirié, Torino
  - ASO SS Antonio e Biagio e Cesare Arrigo, Alessandria
  - Ospedale Oncologico, Bari
  - Policlinico S.Orsola Malpighi, Bologna
  - Spedali Civili, Brescia
  - Ospedale Armando Businco, Cagliari
  - ASO S. Croce e Carle, Cuneo
  - Az. Ospedaliero Universitaria Careggi, Florence
  - IRCCS San Raffaele, Milan
  - Ospedale Cà Granda Niguarda, Milan
  - Univ. Studi Federico II, Napoli
  - ASO Maggiore della Carità Ematologia, Novara
  - Policlinico Monteluce, Perugia
  - Ospedale Bianchi-Melacrino-Morelli, Reggio Calabria
  - Università La sapienza Policlinico Umberto I, Roma
  - Spedali Riuniti, Siena
  - ASO San Giovanni Battista SC Ematologia 2, Torino
  - Policlinico Universitario, Udine